CLINICAL TRIAL: NCT00958828
Title: Clinical Evaluation of Two Daily Disposable Lenses in a Population of Daily Disposable (DD) Lens Wearers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CIBA VISION (Industry)
Responsible Party: Sponsor
Organization: Alcon Research (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: P-337-C-028
Record Dates: First submitted 2009-08-11; First posted 2009-08-13 (Estimated); Results first posted 2010-10-19 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-01

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nelfilcon A / Narafilcon A (Other): Nelfilcon A contact lenses, then Narafilcon A contact lenses
  Interventions: Device: Nelfilcon A contact lens; Device: Narafilcon A contact lens
- Narafilcon A / Nelfilcon A (Other): Narafilcon A contact lenses, then Nelfilcon A contact lenses
  Interventions: Device: Nelfilcon A contact lens; Device: Narafilcon A contact lens

INTERVENTIONS:
Device: Nelfilcon A contact lens — Spherical, soft contact lens for daily disposable wear
Device: Narafilcon A contact lens — Spherical, soft contact lens for daily disposable wear

SUMMARY:
The purpose of this study is to evaluate the performance of two daily disposable contact lenses in a population of daily disposable contact lens wearers.

ELIGIBILITY:
Inclusion Criteria:

* Currently wearing any spherical daily disposable contact lens except the two study products for at least 3 months prior to enrollment.
* Currently wearing contact lenses at least 8 hours/day and 5 days/week.
* Other protocol inclusion/exclusion criteria may apply.

Exclusion Criteria:

* Eye injury or surgery within twelve weeks immediately prior to enrollment.
* Currently enrolled in any clinical trial.
* Prior history of corneal or refractive surgery.
* Monovision correction.
* Other protocol inclusion/exclusion criteria may apply.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2009-07; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

RESULTS

PARTICIPANT FLOW:
Period: Period 1, 1 Week of Wear
Arm/Group | Nelfilcon A / Narafilcon A | Narafilcon A / Nelfilcon A
Started | 89 | 89
Completed | 89 | 88
Not Completed | 0 | 1
Not completed — Randomization break | 0 | 1
Period: Period 2, 1 Week of Wear
Arm/Group | Nelfilcon A / Narafilcon A | Narafilcon A / Nelfilcon A
Started | 89 | 88
Completed | 89 | 87
Not Completed | 0 | 1
Not completed — Unacceptable lens fit | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Overall: This reporting group includes all enrolled and dispensed subjects.
Arm/Group | Overall
Number analyzed (Participants) | 178
Age Continuous [Mean (Standard Deviation); unit: years] | 30.0 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 111
  Male | 67

OUTCOME MEASURES:

1. Primary Outcome: Overall Lens Satisfaction
Description: Overall Lens Satisfaction, as interpreted by the subject and reported by the subject on a questionnaire as a single, retrospective evaluation of 1-week's wear time. Overall lens satisfaction was measured on a 10-point scale, with 1 being poor and 10 being excellent.
Time Frame: After 1 week of wear
Population: Per protocol
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Nelfilcon A Contact Lens | Narafilcon A Contact Lens
Number analyzed (Participants) | 174 | 175
Units on a scale | 7.5 (2.2) | 7.5 (2.3)

ADVERSE EVENTS:
Time Frame: 39 days, duration of the trial
Arm/Group | Nelfilcon A Contact Lens | Narafilcon A Contact Lens
Serious Adverse Events (participants affected / at risk) | 0/177 | 0/178
Other Adverse Events (participants affected / at risk) | 0/177 | 0/178

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
For a period of 10 years, the clinical investigator must hold all trial-related information and documents confidential and must agree to obtain sponsor's written consent before discussing, presenting, publicizing, or otherwise disclosing any preclinical and/or clinical data or impressions from this trial.